CLINICAL TRIAL: NCT04452903
Title: A Communication Enhancing Intervention to Improve Patients' Perception of Physiotherapy Consultations: A Randomized Controlled Trial
Brief Title: A Communication Enhancing Intervention to Improve Patients' Perception of Physiotherapy Consultations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0127-19-com2
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-06

CONDITIONS: Communication
Keywords: communication skills; Consultation reassurance questionnaire
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant (patients of the physiotherapists) are unaware of the intervention.
  The outcome assessor will not know who was in the intervention group and who was in the control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reassurance intervention (Experimental): The physiotherapist in the intervention group (n=15) will participate in a 3-hour communication skill workshop, followed by a month-long period to assimilate and implement the new set of skills, with supervision available by phone from the trainers.
  Interventions: Behavioral: communication skills
- Control (No Intervention): The physiotherapist in the control group (n=15) receives no training.

INTERVENTIONS:
Behavioral: communication skills — 3-hour communication skill workshop, followed by a month-long period to assimilate and implement the new set of skills, with supervision available by phone from the trainers.
  Arms: Reassurance intervention

SUMMARY:
The aim of this study is to test the effectiveness of a single training session in communication skills at improving patients' perceptions of physiotherapy consultations.

DETAILED DESCRIPTION:
Population: Physiotherapists Detail: Physiotherapists (n=30) who work at 'Clalit' institute's (public health management organization in Israel) at four physiotherapy clinics.

Intervention: A single session of training in consultation-based communication skills Detail: a 3-hour communication skill workshop, followed by a month-long period to assimilate and implement the new set of skills, with supervision available by phone from the trainers.

Comparison: No training Detail: The control group receives no extra training. Outcome: New patients' perception of consultations Detail: The Primary Outcome Measure is the Consultation-Based Reassurance Questionnaire (CRQ) The CRQ measures patients' perceptions of consultation. It consists of four subscales, each with three items: data-gathering, relationship-building, generic reassurance, and cognitive reassurance. The investigators are assessing change between two-time points (before and after the intervention). And also, the difference between study groups. This is collected twice: at baseline, and at follow up, from the intervention and control groups.

Type of Question: therapy Detail: The study tests whether a single training sessions can improve communication in consultations with physiotherapists.

Type of Study: RCT

Detail: Stage 1: Pre-randomization:

The physiotherapists (n=30) will hand out a Consultation-Based Reassurance Questionnaire (CRQ) in a sealed envelope to each eligible patient (age 18+) they receive for the first consultation in two weeks period. The patient will complete the questionnaire in private, post consultation, and place it in a closed box. The physiotherapist will recruit a minimum of five patients each (n>150).

Baseline measures are: age, gender, pain area, chronicity, pain severity, disability, satisfaction from the consultation and the Consultation-Based Reassurance Questionnaire.

Stage 2: Randomization:

The process for randomization:

First, participating physiotherapists will be matched for gender, seniority, and quality of reassurance in every clinic. They will then be allocated into one of the two arms at random (1:1), according to a computer random number list.

Stage 3: Follow up:

After the intervention, both the intervention and control groups will again hand out the questionnaires (age, gender, pain area, chronicity, pain severity, disability, satisfaction from the consultation and the CRQ) to new eligible patients that arrive for the first consultation. The physiotherapist will recruit a minimum of ten patients each (total sample therefore n> 300, minimum number per arm=150).

sample size The sample size was calculated with G*Power 3.1.9.4 using the t-test family to detect the difference between two independent means (two groups). The input parameters were as follows: for a two-tailed test, assuming a medium effect size of 0.5, α=0.05, and β=0.95, the total sample size recommended was 210 participants. One hundred five participants in each study group (intervention and control).

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapists:

  * Working for Clalit Health Services. Dan-Petach Tikva region
  * Willing to participate in a 3-hour communication skills workshop
* Patients:

  * over the age of 18
  * literate in Hebrew
  * Willing to participate in the study

Exclusion Criteria:

* Unwilling to participate in the trial
* Illiterate in Hebrew

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Consultation reassurance questionnaire (0-72). Change is being assess before and after the intervention. | measure assessing change between two time points: base line and at two month.
  A questionnaire that measures patients' perceptions of consultation- higher values represent a better communication skills

SECONDARY OUTCOMES:
The numeric pain rating scale (0-10) | 2 month
  For the most severe and average pain intensity ( 0= no pain and 10 =the worst pain)
Disability (0-10) | 2 month
  For disability (0= no disability and 10 =the worst disability)
Satisfaction (0-10) | 2 month
  For satisfaction from the first consultation with the physiotherapist (0= no satisfied at all and 10 =very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Noa Ben Ami, PhD, Principal Investigator — Ariel University
Locations (1):
- Distric DAN - PETACH TIKVA, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holt N, Pincus T. Developing and testing a measure of consultation-based reassurance for people with low back pain in primary care: a cross-sectional study. BMC Musculoskelet Disord. 2016 Jul 12;17:277. doi: 10.1186/s12891-016-1144-2. PMID 27405870
- [Result] Pincus T, Holt N, Vogel S, Underwood M, Savage R, Walsh DA, Taylor SJC. Cognitive and affective reassurance and patient outcomes in primary care: a systematic review. Pain. 2013 Nov;154(11):2407-2416. doi: 10.1016/j.pain.2013.07.019. Epub 2013 Jul 18. PMID 23872104
- [Result] Holt N, Mansell G, Hill JC, Pincus T. Testing a Model of Consultation-based Reassurance and Back Pain Outcomes With Psychological Risk as Moderator: A Prospective Cohort Study. Clin J Pain. 2018 Apr;34(4):339-348. doi: 10.1097/AJP.0000000000000541. PMID 29509169